CLINICAL TRIAL: NCT06316102
Title: Piloting a Multilevel Intervention to Promote Viral Suppression Among Transgender Women Living With HIV in Santo Domingo
Brief Title: Promoting Viral Suppression Among Transgender Women Living With HIV in Santo Domingo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Instituto Dermatológico y Cirugía de Piel (IDCP) (Unknown); George Washington University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-3282; R34MH129218 (NIH)
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-08

CONDITIONS: HIV
Keywords: transgender women; transfeminine people; HIV; Stigma; Cohesion; Multilevel intervention
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group will not receive an intervention; however, provider training in gender affirmation will be conducted at the clinic level, so control participants may be exposed to changes in provider attitudes and practices.
- Gender Affirming Abriendo Puertas (Opening Doors) (GAP) (Experimental): This group will be exposed to all four components of the multilevel intervention.
  1) individual counseling and education; 2) peer navigation; 3) provider capacity building; and 4) community support building.
  Interventions: Behavioral: Gender Affirming Abriendo Puertas (Opening Doors) (GAP)

INTERVENTIONS:
Behavioral: Gender Affirming Abriendo Puertas (Opening Doors) (GAP) — Multilevel intervention with 4 components
  Arms: Gender Affirming Abriendo Puertas (Opening Doors) (GAP)

SUMMARY:
This study includes an adapted multilevel intervention, Abriendo Puertas (Opening Doors), including individual counseling, peer navigation, and community mobilization for transfeminine people living with HIV in the Dominican Republic using an iterative consultation process. Prior to this randomized controlled trial, feasibility and initial effects on HIV care and treatment behaviors were assessed with 30 trans women living with HIV (no control group) and documented positive trends in antiretroviral therapy use (70% to 85%, p=0.03), missed care appointments (35% to 20%, p=0.39) and antiretroviral therapy adherence (86% to 96%, p=0.50). Participants emphasized that trusting intervention staff and being treated with respect in individual sessions allowed them to improve self-esteem. Limited trust and cohesion among trans women, however, inhibited more extensive engagement with peer navigation and community activities. In response, the study team identified two key modifications to strengthen and further tailor the intervention for transfeminine people living with HIV: 1) integrate more gender affirming content, including with providers and 2) focus on building trust among transfeminine people through sequential implementation of individual and then community components. The purpose of the proposed study is to conduct a pilot randomized trial of the Gender-affirming Abriendo Puertas intervention. In Aim 1, the preliminary efficacy of the Gender-affirming Abriendo Puertas intervention on viral suppression among transfeminine people randomized to the intervention compared to those randomized to control will be assessed. The research study will randomly assign transfeminine people living with HIV to the Gender-affirming Abriendo Puertas intervention (n=60) (individual counseling, peer navigation, provider training, and community support building) or control group (n=60). There will be baseline, 6, and 12-month surveys and viral load assessments to assess differences across study arms. In Aim 2, the study team will examine pathways of influence (e.g. decreased stigma, increased cohesion) and experiences with the intervention to identify specific areas for improvement and scale up. Longitudinal qualitative interviews will be conducted at baseline, 6, and 12 months with 20 intervention participants. Together with surveys, the study team will assess how Gender-affirming Abriendo Puertas participation affects pathways between stigma, cohesion, and HIV outcomes. The study team will also elicit experiences and recommendations from providers and intervention staff in focus groups at 6 (n=2) and 12 months (n=2).

ELIGIBILITY:
Inclusion Criteria:

* being at least 18 years of age;
* assigned male at birth but self-identify as transfeminine (using locally appropriate terminology);
* confirmed HIV positive diagnosis using a single rapid test

Exclusion Criteria:

* There is a small group of individuals (approximately 20) who participated in a previous adaptation study to develop the intervention that will be tested in the proposed study. These individuals will not be eligible since they have already been exposed to an earlier version of the intervention.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must have a transfeminine identity.
Enrollment: 121 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Viral Suppression (HIV), 6 months | 6 months
  For viral load assessments of HIV, a 10 mL tube of ethylenediaminetetraacetic acid anti-coagulated blood will be drawn.
  <400 copies/mL= viral suppression >=400 copies/mL=no viral suppression
Viral Suppression (HIV), 1 year | 1 year
  For viral load assessments of HIV, a 10 mL tube of ethylenediaminetetraacetic acid anti-coagulated blood will be drawn.
  <400 copies/mL= viral suppression >=400 copies/mL=no viral suppression
Retention in HIV care, 6 months | 6 months
  Participants who have received HIV care will answer the question:
  In the past 6 months, how many HIV appointments have you missed? 0 = Retention in HIV care >0 = No retention in HIV care
Retention in HIV care, 1 year | 1 year
  Participants who have received HIV care will answer the question:
  In the past 6 months, how many HIV appointments have you missed? 0 = Retention in HIV care >0 = No retention in HIV care
Antiretroviral therapy adherence, 6 months | 6 months
  Participants on antiretroviral therapy will be asked:
  During the last 4 days, how many days did you not take your entire antiretroviral therapy dose? 0 = No antiretroviral therapy interruption >0 = Antiretroviral therapy interruption
Antiretroviral therapy adherence, 1 year | 1 year
  Participants on antiretroviral therapy will be asked:
  During the last 4 days, how many days did you not take your entire antiretroviral therapy dose? 0 = No antiretroviral therapy interruption >0 = Antiretroviral therapy interruption
Antiretroviral therapy interruption, 6 months | 6 months
  Participants on antiretroviral therapy will be asked:
  In the past 6 months, have you stopped or suspended your antiretrovirals?
  No = No antiretroviral therapy interruption Yes = Antiretroviral therapy interruption
Antiretroviral therapy interruption, 1 year | 1 year
  Participants on antiretroviral therapy will be asked:
  In the past 6 months, have you stopped or suspended your antiretrovirals?
  No = No antiretroviral therapy interruption Yes = Antiretroviral therapy interruption

SECONDARY OUTCOMES:
Depression, 6 months | 6 months
  Patient Health Questionnaire-9: 0-9=No depressive symptoms; 10-27=depressive symptoms.
  Response options:
  No day, Several days, More than half the days, Almost every day
  Items about previous 2 weeks:
  You have little interest or pleasure in doing things. You have felt down, depressed, or hopeless. You have had difficulty staying or falling asleep or you have slept too much You have felt tired or with little energy You have had little appetite or have eaten excessively You have felt badly about yourself - or you think you are a failure or that you have done wrong to yourself or your family You have had difficulty concentrating on certain activities, like watching tv or movies You have moved or talked so slowly that other people noticed it You have been so restless or agitated that you have been moving more than normal and others have noticed it You have thought that you would be better off dead or you have thought about harming yourself in some way
Depression, 1 year | 1 year
  Patient Health Questionnaire-9: 0-9=No depressive symptoms; 10-27=depressive symptoms.
  Response options:
  No day, Several days, More than half the days, Almost every day
  Items about previous 2 weeks:
  You have little interest or pleasure in doing things. You have felt down, depressed, or hopeless. You have had difficulty staying or falling asleep or you have slept too much You have felt tired or with little energy You have had little appetite or have eaten excessively You have felt badly about yourself - or you think you are a failure or that you have done wrong to yourself or your family You have had difficulty concentrating on certain activities, like watching tv or movies You have moved or talked so slowly that other people noticed it You have been so restless or agitated that you have been moving more than normal and others have noticed it You have thought that you would be better off dead or you have thought about harming yourself in some way
Anxiety, 6 months | 6 months
  positive screening for anxiety symptoms in the previous 2 weeks. Measured using the Hospital Anxiety and Depression Scale - Anxiety which consists of 7 items.
  Score 0-7 = No anxiety symptoms Score 8-21 = anxiety symptoms
  Items:
  I feel tense or nervous
  * All the times, many times, sometimes, never I have a strange feeling, as if there were butterflies in my stomach
  * Never, on occasion, frequently, very often I have a sense of fear, as if something horrible were going to happen to me
  * Definitely and it is very strong, yes but no too strongly, a little but it doesn't worry me, never I feel restless, as if I couldn't stop moving
  * A lot, a good deal, not much, never My mind is full of worries
  * most of the time, frequently, sometimes but not often, only on occasion Sudden feelings of panic come over me
  * very frequently, often, not often, rarely I can sit comfortably and feel relaxed
  * always, generally, not often, never
Anxiety, 1 year | 1 year
  positive screening for anxiety symptoms in the previous 2 weeks. Measured using the Hospital Anxiety and Depression Scale - Anxiety which consists of 7 items.
  Score 0-7 = No anxiety symptoms Score 8-21 = anxiety symptoms
  Items:
  I feel tense or nervous
  * All the times, many times, sometimes, never I have a strange feeling, as if there were butterflies in my stomach
  * Never, on occasion, frequently, very often I have a sense of fear, as if something horrible were going to happen to me
  * Definitely and it is very strong, yes but no too strongly, a little but it doesn't worry me, never I feel restless, as if I couldn't stop moving
  * A lot, a good deal, not much, never My mind is full of worries
  * most of the time, frequently, sometimes but not often, only on occasion Sudden feelings of panic come over me
  * very frequently, often, not often, rarely I can sit comfortably and feel relaxed
  * always, generally, not often, never
Substance use, 6 months | 6 months
  Yes = used any type of drug in the previous 6 months No = did not use any type of drug in the previous 6 months
Substance use, 1 year | 1 year
  Yes = used any type of drug in the previous 6 months No = did not use any type of drug in the previous 6 months
Binge drinking, 6 months | 6 months
  No = consumes 6+ drinks on one occasion less than once a month Yes = consume 6+ drinks on one occasion at least monthly
Binge drinking, 1 year | 1 year
  No = consumes 6+ drinks on one occasion less than once a month Yes = consume 6+ drinks on one occasion at least monthly
Self-esteem, 6 months | 6 months
  Rosenberg self-esteem scale; analyzed as a continuous variable. A higher score indicates higher self-esteem
  Response options:
  Totally agree = 4 Agree = 3 Disagree = 2 Totally disagree = 1
  Items:
  In general, I am satisfied with myself Sometimes, I think I am not good at anything I feel like I have some good qualities I am capable of doing things as well as the majority of people I feel like I don't have many things to feel proud about Sometimes I feel really useless I feel like I am worth less than most people I wish to respect myself more Definitively, I think I am a failure I have a positive attitude toward myself
  *Items 2, 5, 6, 8, 9 are reverse scored.
Self-esteem, 1 year | 1 year
  Rosenberg self-esteem scale; analyzed as a continuous variable. A higher score indicates higher self-esteem
  Response options:
  Totally agree = 4 Agree = 3 Disagree = 2 Totally disagree = 1
  Items:
  In general, I am satisfied with myself Sometimes, I think I am not good at anything I feel like I have some good qualities I am capable of doing things as well as the majority of people I feel like I don't have many things to feel proud about Sometimes I feel really useless I feel like I am worth less than most people I wish to respect myself more Definitively, I think I am a failure I have a positive attitude toward myself
  *Items 2, 5, 6, 8, 9 are reverse scored.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Barrington, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Instituto Dermatológico y Cirugía de Piel (IDCP), Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2025-10-08): https://cdn.clinicaltrials.gov/large-docs/02/NCT06316102/Prot_002.pdf
  • Statistical Analysis Plan (2024-03-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT06316102/SAP_000.pdf
  • Informed Consent Form (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT06316102/ICF_001.pdf